CLINICAL TRIAL: NCT06071728
Title: Restoring Glycocalyx Thickness in Older Adults to Improve Vascular Function
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Gary L. Pierce, PhD, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202204445
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Aging; Vascular Stiffness; Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocalyx Pro (Active Comparator): Subjects will receive 6 capsules per day (3,712mg) of Endocalyx Pro (Microvascular Health Solutions, US Patent Number: 9943572), a commercially available supplement that includes a proprietary blend of glycocalyx precursors and antioxidants
  Interventions: Dietary Supplement: Endocalyx Pro (Microvascular Health Solutions, US Patent Number: 9943572)
- Placebo (Placebo Comparator): Subjects will ingest placebo pills
  Interventions: Dietary Supplement: Endocalyx Pro (Microvascular Health Solutions, US Patent Number: 9943572)

INTERVENTIONS:
Dietary Supplement: Endocalyx Pro (Microvascular Health Solutions, US Patent Number: 9943572) — Subjects will receive Endocalyx Pro (Microvascular Health Solutions, US Patent Number: 9943572) (3,712mg) or placebo for 12 weeks.

SUMMARY:
The glycocalyx serves as the interface between flowing blood and endothelial cells, the single cell layer that lines blood vessels, and is crucial for normal blood vessel function. Specifically, the glycocalyx protects endothelial cells from oxidative stress and inflammation and enables blood vessel dilation, which is largely dependent on the bioavailability of the vasodilatory molecule nitric oxide. Importantly, glycocalyx thickness decreases with age and is predictive of major adverse cardiovascular events in older adults free of cardiovascular disease. Therefore, interventions aimed at restoring glycocalyx thickness in older adults are desperately needed. Endocalyx Pro is a commercially available glycocalyx precursor supplement, manufactured by Microvascular Health Solutions, designed to 1) repair a damaged glycocalyx, 2) protect against damage to the glycocalyx, and 3) synthesize new glycocalyx components, and has been used to increase glycocalyx thickness in humans. However, no study has tested if glycocalyx thickness restores glycocalyx thickness in older adults and improves blood vessel function. Thus, the purpose of this investigation is to determine if 12-weeks of Endocalyx Pro supplementation alters glycocalyx thickness and blood vessel function in older adults. The investigators will use a camera placed under the tongue to determine glycocalyx thickness. The investigators will measure blood vessel function by measuring brachial artery dilation with ultrasound and arterial stiffness using pressure probes placed on the carotid and femoral artery.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85 years
* Able to undergo cardiovascular testing procedures including fasting overnight and holding selected morning medication doses.
* Ability to understand and willingness to sign a written informed consent document.
* Ability to lie comfortably for up to 90 minutes
* Women only: Post-menopausal

Exclusion Criteria:

* Current or history of CVD disease (heart attack, stroke, heart failure, cardiomyopathy or peripheral artery disease, heart angioplasty/stent or bypass surgery, valve replacement, carotid endarterectomy, heart transplant.
* Medical history of stroke or other neurological disorder or systemic illness that could potentially affect cognition or brain function (outside of a diagnosis of MCI, Alzheimer's Disease) or could affect their safety or comfort while undergoing the imaging or cardiovascular studies.
* Subjects with evidence of cardiovascular disease at baseline or during the exercise test (evidence of myocardial infarction, abnormal cardiac arrhythmia, myocardial ischemia, conduction delays, >1mm ST segment depression or elevation; >3 beat ventricular tachycardia; atrial fibrillation) will be excluded from the study.
* Wilson's disease, hemochromatosis
* Individuals taking clonidine or other short-acting beta blocker
* Resting blood pressure > 149 mmHg systolic and/or 99mmHg diastolic
* BMI > 40 kg/m2
* Medical history of chronic major psychiatric or current diagnosis of major psychiatric disease (other than dementia).
* Unable to provide informed consent due to cognitive impairment
* Current clinically abnormal thyroid function not adequately regulated by thyroid hormone supplementation or medication.
* Allergic to olives, artichokes, grapes or melons
* Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, hookah, electronic cigarettes) or living with someone who smokes/has smoked in the past 3 months.
* Current diagnosis of diabetes (Type I or insulin dependent Type II)
* Current diagnosis of COPD, cystic fibrosis, emphysema, chronic bronchitis
* History of renal failure, dialysis or kidney transplant
* Current diagnosis or history of liver disease or HIV/AIDS, or cancer requiring chemotherapy or radiation.
* Current diagnosis or history of rheumatoid arthritis, systemic lupus erythematosus, Wegener's granuomatosis
* Vulnerable populations (prisoners, etc) will not be eligible.
* Unwillingness to wash out from a vitamin or dietary supplement regime prior to enrollment and maintain throughout the duration of the study.
* Inability to comply with experimental instructions.
* Uncontrolled intercurrent illness that would limit compliance with study requirements per investigator.
* Inability to fast or hold morning medications doses until after testing is complete.
* Hormone replacement use within the past 6 months
* Currently enrolled in another study using an study medication, supplement, device or intervention.
* Initiation of a new prescription medication or change in dose/frequency in the past three months. Individuals will be become eligible after the medication/dose/frequency has been stable for 3 months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation (FMD) | Baseline and 12 weeks
  Conduit artery vascular endothelial function
Perfused boundary region (PBR) | Baseline and 12 weeks
  Microvascular endothelial glycocalyx thickness

CONTACTS AND LOCATIONS:
Overall Officials: Gary Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Individual deidentified data will be shared with other researchers upon reasonable request.